CLINICAL TRIAL: NCT03884946
Title: Getting Off: : A Theory-based mHealth Intervention for Methamphetamine-using MSM
Brief Title: The Getting Off App for Methamphetamine-Using Gay and Bisexual Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA045562 (NIH); R01DA045562 (NIH)
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-03

CONDITIONS: Methamphetamine Abuse; HIV/AIDS
Keywords: MSM; mHealth; App
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Two randomly assigned arms will receive the same intervention (i.e., an app) at staggered intervals. At the end of one month, participants in the immediate arm will have received the app, but participants in the delayed arm will not. At this point, the two groups represent an RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Delivery (Active Comparator): Participants randomized into the Immediate Delivery arm (n = 113) receive access to the app immediately upon enrollment, and are given a pre- (baseline) and post- (one month post-baseline) test.
  Interventions: Other: Getting Off App
- Delayed Delivery (Placebo Comparator): Participants randomized into the Delayed Delivery arm (n = 113) don't receive access to the app until one month post-baseline. For the RCT portion of the analysis, they will also be assessed at baseline and one month post-baseline (i.e., a pre- and post- prior to app exposure, making them the placebo comparator).
  Interventions: Other: Getting Off App

INTERVENTIONS:
Other: Getting Off App — A mobile phone application based on the "Getting Off" methamphetamine treatment manual. Participants download the app and progress through the sessions of the Getting Off intervention through the administration of games, activities, lessons, quizzes, and tutorials. There are 24 sessions total in the app, each addressing a different component of the methamphetamine treatment process. The fundamental basis of the app is gay-specific cognitive behavioral therapy, with elements of motivational interviewing, social support theory, and health belief model dynamics included.

SUMMARY:
A commonly used manualized outpatient methamphetamine intervention for gay and bisexual men, "Getting Off," is being translated into a mobile phone application (i.e., app) available for download through common app marketplaces. The application will provide games, guided lessons, informational support, and resources to gay and bisexual men seeking to reduce their methamphetamine use and risky sexual behaviors.

DETAILED DESCRIPTION:
The research team will conduct formative research to translate the 24 Getting Off sessions from a group-based manual-driven intervention to a computerized app, conduct alpha phase post-development bug testing, conduct beta phase usability pilot testing, and refine the app according to alpha- and beta-phase testing. Four focus groups will provide input on the development of the Getting Off app (further input will be obtained through an ongoing Consumer Advisory Board and usability pilot testing) with: 1) out-of-treatment, methamphetamine-using MSM (n=~8); 2) methamphetamine-using men who have sex with men (MSM) who are currently in outpatient treatment in the brick-and-mortar Getting Off program at the study site (n=~8); 3) prior methamphetamine-using MSM with a minimum of one year recovery who have completed a minimum 18/24 sessions (75%) of the brick-and-mortar Getting Off program; and, 4) prior methamphetamine-using MSM with a minimum of one year recovery who have had no previous experience or knowledge of the Getting Off intervention (n=~8). The focus groups will be structured to provide guidance on translating Getting Off into an app that is responsive to culture (e.g., sexuality; HIV prevention/care including pre-exposure prophylaxis (PrEP) uptake, adherence and persistence, antiretroviral therapy (ART) adherence, viral load suppression) and methamphetamine treatment needs.

Following app development, and to ensure benchmarks have been met, alpha phase testing will uncover and remove unwanted bugs, and beta phase usability pilot testing will be conducted with members of the target population (N=30) to test the feasibility, acceptability, and preliminary effects of the Getting Off app. Furthermore, the pilot testing will be utilized to ensure the functionality of the app (i.e., that the app is user-friendly and all features function appropriately).

Behavioral assessments will be conducted at baseline and at 1-month follow-up.

The study team will then conduct a randomized controlled trial (RCT) to evaluate reductions of methamphetamine use and HIV sexual risk behaviors, and increased advancement along the HIV Prevention or Care Continuum, using three approaches: a) two-arm RCT to determine intervention effects through comparison of the immediate delivery (ID; n=150) and delayed delivery (DD; n=150) arms; b) an observed treatment effects analysis powered for prospective sub-group to compare longitudinal pre/post data from the pooled ID and DD arms (N=300); and, c) a two-arm historical matched comparison design to evaluate the outcomes of the Getting Off app (ID+DD; N=300) relative to a matched sample of participants having previously attended the brick-and-mortar group-based Getting Off intervention (N~600; total N=900).

Following screening, informed consent and baseline assessments, participants will be randomized into one of two arms: Arm A: Immediate access to the Getting Off app (ID); or, Arm B: Participants will have access to the Getting Off app after a delayed 30-day period (DD). Participants in both arms will receive the same Getting Off app and participants in both arms will be given 30-days to engage with the app. The randomized two-arm repeated measures design will assess participants at 1-, 2- (DD arm only), 3-, 6-, and 9-months post-randomization to determine longitudinal intervention effects, observed treatment effects, and a historical comparison with a matched sample of participants who have attended the brick-and-mortar group-based Getting Off intervention.

ELIGIBILITY:
Inclusion Criteria:

Self-identified man who has sex with men (MSM) Any methamphetamine use in the past 365 days Between the ages of 18-65 years Able and willing to provide informed consent.

Exclusion Criteria:

Did not identify as a man who had sex with a man No methamphetamine use in the past 365 days Younger than 18 or older than 65 years Not able or willing to provide informed consent.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Reback, Ph.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Community Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share IPD.

REFERENCES:
- [Derived] Reback CJ, Fletcher JB, Mata RP. A Theory-Based mHealth Intervention (Getting Off) for Methamphetamine-Using Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Feb 22;10(2):e22572. doi: 10.2196/22572. PMID 33616547

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Delivery (ID; n=113): Getting Off is a 24-session Cognitive Behavioral Therapy (CBT) intervention specifically designed to intervene on the intersectionality of methamphetamine use and concomitant sexual risk behaviors among SMM, and to increase advancement along the HIV prevention and care continua. Critical CBT skills within Getting Off include, for example, education on internal and external triggers, thought stopping, relapse prevention, relapse analysis including the identification of emotional states that can signal relapse, and the adoption of prosocial and healthy behaviors. All sessions are embedded within the specific cultural, social, and sexual components of methamphetamine use among SMM. Throughout the 24 sessions, equal content is given to the reduction of methamphetamine use and sexual risk behaviors.
- Delayed Delivery (DD; n=113): The participants in the DD group received the same intervention as those in the ID group, but after a 30-day delayed period.
Period: Overall Study
Arm/Group | Immediate Delivery (ID; n=113) | Delayed Delivery (DD; n=113)
Started | 113 | 113
Completed | 85 | 94
Not Completed | 28 | 19

BASELINE CHARACTERISTICS:
Groups:
- Immediate Delivery: Getting Off is a 24-session Cognitive Behavioral Therapy (CBT) intervention specifically designed to intervene on the intersectionality of methamphetamine use and concomitant sexual risk behaviors among SMM, and to increase advancement along the HIV prevention and care continua. Critical CBT skills within Getting Off include, for example, education on internal and external triggers, thought stopping, relapse prevention, relapse analysis including the identification of emotional states that can signal relapse, and the adoption of prosocial and healthy behaviors. All sessions are embedded within the specific cultural, social, and sexual components of methamphetamine use among SMM. Throughout the 24 sessions, equal content is given to the reduction of methamphetamine use and sexual risk behaviors.
- Delayed Delivery: The Delayed Delivery group received the exact same Getting Off app, but after a 30-day delay.
- Total: Total of all reporting groups
Arm/Group | Immediate Delivery | Delayed Delivery | Total
Number analyzed (Participants) | 113 | 113 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (9.5) | 45.3 (10.3) | 45.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 113 | 113 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 37 | 77
  Not Hispanic or Latino | 63 | 67 | 130
  Unknown or Not Reported | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 27 | 29 | 56
  White | 52 | 44 | 96
  More than one race | 11 | 11 | 22
  Unknown or Not Reported | 20 | 24 | 44
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 113 | 113 | 226
Baseline Methamphetamine Use [Mean (Standard Deviation); unit: days] | 13.6 (11.3) | 14.5 (11.8) | 14.4 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Use
Description: Days of participant self-reported methamphetamine use in the past 30 days.
Time Frame: from baseline to 9-months post randomization
Population: Gay and bisexual men that use methamphetamine
Measure: Mean (Standard Deviation); unit: days
Groups:
- Immediate Delivery (ID): Participants who were randomized into the ID condition were immediately given a unique user passcode to access the intervention app
- Delayed Delivery (DD): Participants who were randomized into the DD arm received their unique user passcode 30 days post-randomization
Arm/Group | Immediate Delivery (ID) | Delayed Delivery (DD)
Number analyzed (Participants) | 113 | 113
days
  Baseline | 13.6 (11.3) | 15.3 (11.2)
  1 month: number analyzed (Participants) | 97 | 95
  1 month | 10.9 (10.3) | 14.5 (11.8)
  2 months: number analyzed (Participants) | 0 | 92
  2 months |  | 14.4 (10.7)
  3 months: number analyzed (Participants) | 81 | 96
  3 months | 9.4 (10.0) | 13.4 (11.6)
  6 months: number analyzed (Participants) | 90 | 90
  6 months | 10.2 (10.7) | 13.2 (11.6)
  9 months: number analyzed (Participants) | 85 | 94
  9 months | 8.8 (9.6) | 11.7 (11.5)

2. Primary Outcome: Methamphetamine Injection
Description: Days participants self-reported methamphetamine injection use in past 30 days
Time Frame: From baseline to 9-months post randomization
Population: gay and bisexual men that use methamphetamine
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Immediate Delivery (ID) | Delayed Delivery (DD)
Number analyzed (Participants) | 113 | 113
days
  Baseline | 2.2 (5.5) | 2.3 (5.9)
  1 month: number analyzed (Participants) | 97 | 95
  1 month | 1.2 (4.4) | 2.3 (5.8)
  2 months: number analyzed (Participants) | 0 | 92
  2 months |  | 2.4 (6.1)
  3 months: number analyzed (Participants) | 81 | 96
  3 months | 0.7 (2.8) | 1.6 (4.6)
  6 months: number analyzed (Participants) | 90 | 90
  6 months | 1.3 (4.7) | 1.6 (5.4)
  9 months: number analyzed (Participants) | 85 | 94
  9 months | 0.8 (2.9) | 0.8 (3.4)

3. Primary Outcome: Condomless Anal Intercourse
Description: Reporting condomless anal intercourse in the past 30 days (yes/no)
Time Frame: baseline to 9-months post randomization
Population: gay and bisexual men that use methamphetamine
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Delivery (ID) | Delayed Delivery (DD)
Number analyzed (Participants) | 113 | 113
Participants
  Baseline | 63 | 54
  1 month: number analyzed (Participants) | 97 | 95
  1 month | 40 | 55
  2 months: number analyzed (Participants) | 0 | 92
  2 months |  | 36
  3 months: number analyzed (Participants) | 81 | 96
  3 months | 32 | 36
  6 months: number analyzed (Participants) | 90 | 90
  6 months | 38 | 35
  9 months: number analyzed (Participants) | 85 | 94
  9 months | 40 | 32

4. Primary Outcome: Condomless Anal Intercourse While High on Methamphetamine
Description: Reporting condomless anal intercourse while high on methamphetamine in the past 30 days (yes/no)
Time Frame: 9-months post randomization
Population: gay and bisexual men that use methamphetamine
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Delivery (ID) | Delayed Delivery (DD)
Number analyzed (Participants) | 113 | 113
Participants
  Baseline | 56 | 49
  1 month: number analyzed (Participants) | 97 | 95
  1 month | 30 | 42
  2 months: number analyzed (Participants) | 0 | 92
  2 months |  | 30
  3 months: number analyzed (Participants) | 81 | 96
  3 months | 26 | 32
  6 months: number analyzed (Participants) | 90 | 90
  6 months | 26 | 28
  9 months: number analyzed (Participants) | 85 | 94
  9 months | 26 | 23

5. Secondary Outcome: ART Initiation
Description: Starting to receive ART among HIV sero-positive participants who were not on ART at baseline (yes/no)
Time Frame: 9-months post randomization
Population: gay and bisexual men that use methamphetamine
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Delivery (ID) | Delayed Delivery (DD)
Number analyzed (Participants) | 15 | 16
Participants | 2 | 5

6. Secondary Outcome: PrEP Initiation
Description: Starting to receive PrEP among HIV sero-negative participants who were not on PrEP at baseline (Yes/No)
Time Frame: 9-months post randomization
Population: gay and bisexual men that use methamphetamine
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Delivery (ID) | Delayed Delivery (DD)
Number analyzed (Participants) | 34 | 37
Participants | 4 | 7

ADVERSE EVENTS:
Time Frame: Up to 9 months post randomization
Description: The definition of adverse event and serious adverse event is the same as clinicaltrials.gov.
Groups:
- Immediate Delivery: Those in the ID arm received access to the app immediately.
- Delayed Delivery: Those in the DD arm received access to the app after 30 days.
Arm/Group | Immediate Delivery | Delayed Delivery
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/113
Other Adverse Events (participants affected / at risk) | 0/113 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT03884946/Prot_SAP_003.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT03884946/ICF_002.pdf